CLINICAL TRIAL: NCT05727982
Title: Identification of Molecular Mechanisms of Coronary Instability in Homogeneous Subsets of Patients With Acute Coronary Syndromes for the Implementation of Precision Medicine (PRECISION Study)
Brief Title: Identification of Molecular Mechanisms of Coronary Instability in Homogeneous Subsets of Patients With Acute Coronary Syndromes for the Implementation of Precision Medicine
Acronym: PRECISION
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Liuzzo Giovanna, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 2747
Record Dates: First submitted 2023-02-02; First posted 2023-02-14 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Acute Coronary Syndrome; Chronic Coronary Syndrome
Keywords: Atherosclerotic plaque; Optical Coherence Tomography
MeSH Terms: conditions — Acute Coronary Syndrome; Plaque, Atherosclerotic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Stool sample for the study of the composition of the intestinal bacterial flora (microbiota) faeces sample can also be collected at home, keeping it at +4°C. Such sample must be transported cold, +4°C, and delivered to the staff within 24 hours polyclinic.
  A venous blood sample of 18cc which will be used to evaluate: 1) the inflammatory profile systemically by measuring the following plasma biomarkers: zonulin, C-reactive protein, IL-1, IL-1Ra, IL-5, IL-6, IL-7, IL-8, IL-9, IL-12, IL-17, IFN-γ, MIP-1b, VEGF, MCP-1 and IL-8, IL-10, TNF- a, TGF-b, LPS, 2) plasma metabolites.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- NSTEMI patients: Patients no ST-segment elevation myocardial infarction (NSTEMI)
  Interventions: Diagnostic Test: Venous blood samples, Biological samples analysis, Cardiology visit.
- SA patients: Patients with Stable Angina (SA) diagnosis
  Interventions: Diagnostic Test: Venous blood samples, Biological samples analysis, Cardiology visit.
- MVD patients: Patients with consecutive Mitral Valve Disease patients (MVD)
  Interventions: Diagnostic Test: Venous blood samples, Biological samples analysis, Cardiology visit.

INTERVENTIONS:
Diagnostic Test: Venous blood samples, Biological samples analysis, Cardiology visit. — These interventions are important to study all patients recruited

SUMMARY:
To further improve the outcome of ACS it is strongly needed to identify new therapeutic targets. This is possible only by improving our knowledge of the multiple molecular mechanisms leading to coronary instability through several pathways. The goal of this project is to define the molecular mechanisms responsible for the four different presentations of ACS, to identify biomarkers for their noninvasive identification and potential new therapeutic targets, thus promoting precision medicine.

DETAILED DESCRIPTION:
This is a multicenter prospective observational study, involving 5 Research Units (RU), the enrollment-phase will take 18 months (month 6 to 24). This is an explorative project that will prospectively enroll: 1) Consecutive patients with an admission diagnosis of ACS with Non ST elevation myocardial infarction (NSTEMI) confirmed at coronary angiography, undergoing OCT evaluation of the culprit coronary plaque before stent implantation for clinical reasons and with a clearly identifiable feature of the culprit plaques according to current European guidelines. ECG changes may include transient ST- segment elevation, persistent or transient ST-segment depression, T-wave inversion, flat T waves or pseudo- normalization of T waves or the ECG may be normal. Taking into account our previous studies, the investigators estimated that between 30-35% of NSTEMI patients will undergo OCT evaluation; 2) Consecutive patients with symptoms of Stable Angina (SA) lasting >12 months, angiographically confirmed coronary artery disease, without any episode suggestive of previous acute event, and no overt ischemic episodes during the last 48 hours, according to current European guidelines. Myocardial ischemia was documented by afunctional test (ie, exercise treadmill testing and/or myocardial perfusion imaging). Patients showing Q waves on 12-lead electrocardiogram and/or abnormal echocardiogram (ie, left ventricular ejection fraction <40% and/or wall motion abnormalities) were excluded. NSTEMI (within 12 hours of symptom onset) and SA patients will be enrolled at the time of their admission to the Coronary Care Unit and to the SubIntensive Cardiac Care Unit, of wich Prof. Giovanna Liuzzo (project PI) is the supervising physician; 3) In the same period, consecutive Mitral Valve Disease patients (MVD) with angiographically normal coronary arteries undergoing surgery for mitral valve regurgitation, age and sex matched 1:3 with NSTEMI patients, will be enrolled as control group. MVD patients will be enrolled at Cardiosurgery Operative Unit, lead by Professor Massimo Massetti.

Our RU1 will enroll:

1. 150 consecutive patients with an admission diagnosis of NSTEMI.
2. 50 consecutive patients with a diagnosis of SA.
3. 50 consecutive MVD.

ELIGIBILITY:
Inclusion Criteria:

* Men and post-menopause women of age 45-80 years; ability to understand and sign the informed consent;
* For NSTEMI and SA patients inclusion criteria will include evidence of obstructive atherosclerosis (> 70% stenosis) at invasive coronary angiography;

Exclusion Criteria:

* Evidence of inflammatory or infectious diseases, malignancies, immunological or haematological disorders;
* Ejection fraction less than 40%;
* Treatment with anti-inflammatory drugs other than low-dose aspirin, and with antibiotic therapies until 1 month before the enrollment.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Patients with plaque rupture and inflammation;
  2. Patients with plaque rupture without inflammation;
  3. Patients with intact fibrous plaque with evidence of thrombus (plaque erosion);
  4. Patients with a smooth plaque.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-09-13 (Actual); Primary Completion 2023-09-05 (Estimated); Study Completion 2024-09-13 (Estimated)

PRIMARY OUTCOMES:
Identify homogeneous subsets of ACS patients at OCT interrogation of the culprit plaque | 2 week
  Using Optical Coherence Tomography

SECONDARY OUTCOMES:
Assess the role of shear stress in coronary instability | 1 year
  On OCT-based reconstruction of coronary lesions and fluid dynamics studies;
Establish the most efficient and cost-effective biomarker panel | 1 years
  Establish the most efficient and cost-effective biomarker panel for the identification of homogeneous ACS patient subsets, this approach is relevant especially in centers where OCT is not available and unravel specific mechanisms and players of coronary instability and to identify molecular therapeutic targets, taking advantage of newomics technologies.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Gemelli, Roma, Italy

IPD SHARING:
Plan to Share IPD: No